CLINICAL TRIAL: NCT00388791
Title: Comparison of Systane Free vs. Saline in the Treatment of Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-S4507
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Dry Eye
Keywords: symptomatology; Schein questionnaire; fluoresceien staining
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Drug: Systane Free

SUMMARY:
The purpose of this study is to compare the efficacy of Systane Free to Saline in decreasing the symptoms of dry eye after aggressive therapy. As a principal outcome measure, we are using the modified Schein dry eye symptomatology questionaire to determine whether any improvement in signs is mirrored by improvement in the Schein Score. Up to 30 dry eye subjects will be dosed six times per day for one month. The typical clinical signs will be onmitored (e.g., corneal staining) along with dyrness symptoms. The hypothesis is that an optimized drop, Systane Free, will be more effective than saline solution in improving dry eye signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

The informed consent document must be read, signed and dated by the subject or legally authorized representative before conducting any procedures. Additionally, the informed consent document must be signed and dated by the individual obtaining consent of the subject.

Adult subjects with mild to moderate dry eye. Criteria for the diagnosis must include two of the three following characteristics as demonstrated at the Eligibility Visit:

Composite symptom score of greater than or equal to 7 on the Schein Questionnaire.

Sodium Fluorescein (NaFl) Tear Break-Up Time less than 7 seconds in both eyes. Cumulative Sodium Fluorescein Corneal Staining greater than or equal to 4 in both eyes on a 0 to 20 point scale.

Rose Bengal corneal staining greater than 4 of 24 maximum for 6 zones. Able and willing to follow study instructions. Subjects must have best corrected visual acuity of twenty twenty five or better in each eye.

The informed consent document must be read, signed and dated by the subject or legally authorized representative before conducting any procedures. Additionally, the informed consent document must be signed and dated by the individual obtaining consent of the subject.

Adult subjects with mild-to-moderate dry eye. Criteria for the diagnosis must include two of the three following characteristics as demonstrated at the Eligibility Visit

Composite symptom score of greater than or equal to 7 on the Schein Questionnaire.

Sodium FluoresceinTear Break-Up Time less than or equal to 7 seconds in both eyes.

Cumulative Sodium Fluorescein Corneal Staining greater than or equal to 4 in both eyes on a 0 to 20 point scale.

Rose Bengal corneal staining greater than 4 of 24 maximum for 6 zones. Able and willing to follow study instructions. Subjects must have best corrected visual acuity of twenty twenty five or better in each eye.

Exclusion Criteria:

History or evidence of ocular or intraocular surgery in either eye within the past six months. LASIK and other keratorefractive procedure patients may participate if the surgery was earlier than 12 months at the time of the beginning of the study.

History or evidence of serious ocular trauma in either eye within the past six months.

History of hypersensitivity to any component of the study medications. These include the artificial tear and the diagnostic dye sodium fluorescein.

History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia, active or recent varicella, viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal disease of the eye.

Use of topical ocular medications during the study period. Subjects using systemic steroids, immunosuppressive agents and/or anti-cholinergics (e.g. cold and allergy medications, tricyclic antidepressants) for treatment of autoimmune connective tissue disease may not be enrolled in the study if they have not been on a stable dosing regimen for a minimum of 30 days prior to the Eligibility Visit. In addition, the dosing regimen must remain stable throughout the 4-week treatment period.

Ocular conditions such as active acute conjunctival infections or iritis. Individuals unwilling to discontinue contact lens wear for seven days prior to the study and throughout the study.

Participation in an investigational drug or device study within 30 days of entering this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Ocular health measures, including corneal staining and rose bengal staining
Symptom scores using the Schein questionnaire
Tear breakup time

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Paugh, Study Director — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California Colleg of Optometry, Fullerton, California, United States